CLINICAL TRIAL: NCT05604469
Title: The Role of Skin Microbiota in Patients With Hepatic or Renal Pruritus
Brief Title: The Role of Skin Microbiota in Hepatic or Renal Pruritus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Essam, Lecturer of Dermatology, Zagazig University
Other Study IDs: 9802-11-10-2022
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Renal Failure; Hepatic Failure; Pruritus
MeSH Terms: conditions — Renal Insufficiency; Liver Failure; Pruritus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A (liver faluire patients with pruritus): Patients with hepatic illness (autoimmune liver diseases, chronic viral hepatitis, and drug-induced liver injury)
  Interventions: Diagnostic Test: Isolation of skin microbiota
- Group B (liver faluire patients without pruritus): Patients with hepatic illness (autoimmune liver diseases, chronic viral hepatitis, and drug-induced liver injury)
  Interventions: Diagnostic Test: Isolation of skin microbiota
- Group C (renal faluire patients with pruritus)
  Interventions: Diagnostic Test: Isolation of skin microbiota
- Group D (renal faluire patients without pruritus)
  Interventions: Diagnostic Test: Isolation of skin microbiota

INTERVENTIONS:
Diagnostic Test: Isolation of skin microbiota — Isolation of skin microbiota including, Staphylococcus epidermidis, Propionibacterium acnes, Pseudomonas aeruginosa, Staphylococcus aureus, Streptococcus pyogenes and Candida.

SUMMARY:
* Various neurotransmitters may share in the pathogenesis of hepatic and renal itching.
* Skin microbiota may share in the pathogenesis of pruritus.

DETAILED DESCRIPTION:
Uremic pruritus (UP) is a frequent phenomenon and it is regarded as one of the most bothersome symptoms in patients with chronic renal disease. The prevalence of UP is still high and reported in around 40% to 50%. UP has an important impact on patients' quality of life and sleep, depression, and increased mortality. The pathogenesis of UP remains blurry, although many different factors have been indicated in the etiology of this symptom, including increased systemic inflammation, abnormal serum parathyroid hormone, calcium, and phosphorus levels, an imbalance in opiate receptors, a neuropathic process, or even skin dryness. This is why until now there is no specific treatment for patients with UP and many of the available therapeutic modalities are not satisfactory Pruritus in liver diseases can often be a debilitating symptom causing significant impairment in quality of life. Not all patients with liver disease develop pruritus and its prevalence varies depending on the underlying cause of liver disease. It is more common in conditions characterized by bile duct inflammatory destruction than in those characterized by hepatocellular injury.

Cutaneous microbiota delivers a diverse and far-reaching influence on our physiology by calling upon the host nervous system. Bacteria make metabolites, toxins, and structural components that are recognized by peripheral and central neurons via matching receptors. Microbiota also indirectly affects neural function by causing endocrine (i.e., keratinocytes) and immune cells to transmit signals (i.e., cytokines, proteases). Itch is a prototypic sensory neural function, and the microbiota propels the itch-scratch cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes. Patients with hepatic illness (autoimmune liver diseases, chronic viral hepatitis, and drug-induced liver injury) or Patients with renal failure Willing to sign an informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sexes. Patients with hepatic illness (autoimmune liver diseases, chronic viral hepatitis, and drug-induced liver injury) or Patients with renal failure Willing to sign an informed consent.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the possible change of skin microbiota in patients with renal or hepatic pruritus | 8 weeks
  Isolation of skin microbiota including, Staphylococcus epidermidis, Propionibacterium acnes, Pseudomonas aeruginosa, Staphylococcus aureus, Streptococcus pyogenes and Candida.

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Essam, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szepietowski JC, Salomon J. Uremic pruritus: still an important clinical problem. J Am Acad Dermatol. 2004 Nov;51(5):842-3. doi: 10.1016/j.jaad.2004.04.003. No abstract available. PMID 15523377
- [Background] Szepietowski JC, Sikora M, Kusztal M, Salomon J, Magott M, Szepietowski T. Uremic pruritus: a clinical study of maintenance hemodialysis patients. J Dermatol. 2002 Oct;29(10):621-7. doi: 10.1111/j.1346-8138.2002.tb00191.x. PMID 12432992
- [Background] Combs SA, Teixeira JP, Germain MJ. Pruritus in Kidney Disease. Semin Nephrol. 2015 Jul;35(4):383-91. doi: 10.1016/j.semnephrol.2015.06.009. PMID 26355256
- [Background] N. V. Bergasa. Frontiers in neuroscience pruritus of cholestasis. In: Carstens E, Akiyama T, editors. Itch: mechanisms and treatment. Boca Raton, FL: CRC Press/Taylor & Francis Group; 2014.
- [Background] Kim HS, Yosipovitch G. The Skin Microbiota and Itch: Is There a Link? J Clin Med. 2020 Apr 22;9(4):1190. doi: 10.3390/jcm9041190. PMID 32331207